CLINICAL TRIAL: NCT05128175
Title: An Open-label, Balanced, Randomized, Five-treatment, Five-period, Five-sequence, Multiple Oral Dose, Crossover Comparative Bioavailability Study of Different Strengths of Carbidopa/Levodopa Extended-release Tablets With Carbidopa and Levodopa Tablets in Normal, Healthy Adult Human Subjects Under Fasting and Fed Conditions
Brief Title: Comparative Bioavailability Study of Carbidopa/Levodopa Extended-Release Tablets Under Fasting and Fed Conditions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai WD Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WD-1603-1005
Record Dates: First submitted 2021-10-27; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-10

CONDITIONS: Parkinson Disease
Keywords: WD-1603; Carbidopa-Levodopa Extended-Release Tablets
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 25 mg /100 mg treatment A group (Experimental): Treatment A: carbidopa/levodopa (25 mg /100 mg)
  Interventions: Drug: WD-1603 Carbidopa-Levodopa Extended-Release Tablets
- 25 mg /150 mg treatment B group (Experimental): Treatment B: carbidopa/levodopa (25 mg/150mg)
  Interventions: Drug: WD-1603 Carbidopa-Levodopa Extended-Release Tablets
- 25 mg /150 mg treatment C group (Experimental): Treatment C: carbidopa/levodopa (25 mg /150 mg)
  Interventions: Drug: WD-1603 Carbidopa-Levodopa Extended-Release Tablets
- 25 mg /150 mg treatment D group (Experimental): Treatment D: carbidopa/levodopa (25 mg /150 mg)
  Interventions: Drug: WD-1603 Carbidopa-Levodopa Extended-Release Tablets
- 25 mg /100 mg placebo group (Placebo Comparator): Treatment E(Reference): Carbidopa and Levodopa tablets (a generic version of Sinemet® IR) 25 mg/100 mg
  Interventions: Drug: WD-1603 Carbidopa-Levodopa Extended-Release Tablets

INTERVENTIONS:
Drug: WD-1603 Carbidopa-Levodopa Extended-Release Tablets — For fasting conditions in the morning, a single oral dose will be administered to each subject under fasting conditions before 5 minutes of serving a standardized vegetarian breakfast as per the randomization schedule; for fasting conditions in the afternoon and evening, a single oral dose will be administered to each subject under fasting condition before 5 minutes of serving standardized vegetarian lunch and dinner as per randomization schedule. For fed condition, single oral dose will be administered to each subject after 30 minutes of serving standardized vegetarian breakfast, lunch and dinner as per randomization schedule. Dosing interval between two subsequent dosing should be 5 hours in each period. There will be one tablet for A, B, C, D and E.
  Other Names: WD-1603

SUMMARY:
It is an open-label, balanced, randomized, five-treatment, five-period, five-sequence, multiple oral dose, crossover comparative bioavailability study of different strengths of carbidopa/levodopa extended-release tablets with carbidopa and levodopa tablets in normal, healthy adult human subjects under fasting and fed conditions. The primary objective of the study is to compare the pharmacokinetic profiles between WD-1603 extended-release formulations and carbidopa and levodopa tablets 25mg/100mg following three times a day after oral administration in fasting and fed conditions in healthy subjects and to compare relative bioavailability between treatments.

DETAILED DESCRIPTION:
Study WD-1603-1005 is to compare the fluctuation index between WD-1603 extended-release formulations and Carbidopa and Levodopa Tablets following three times a day oral administration and the food effect on the initial absorption of levodopa in the morning in healthy subjects. At least 15 subjects will be enrolled at the beginning of the study and the order of receiving the Treatment A, B, C, D & E for each subject during all the periods of the the study will be determined according to a randomization schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Normal, healthy adult human volunteers between 18 to 45 years of age (both inclusive).
2. Having a Body Mass Index (BMI) between 18.5 to 29.9 (both inclusive), calculated as weight in kg/ height in m2, a minimum body weight of 50.0 kg.
3. Not having any significant disease or clinically significant abnormal findings during screening, medical history, clinical examination, laboratory evaluations, 12- lead ECG, and X-ray chest (P/A view) recordings.
4. In the case of female subjects:

a. Surgically sterilized at least 6 months prior to study participation or If of childbearing potential is willing to use a suitable and effective double barrier contraceptive method or intra-uterine device during the study and for at least 28 days after the last study drug administration.

And b. Serum Pregnancy test must be negative.

Exclusion Criteria:

1. Known hypersensitivity or idiosyncratic reaction to Carbidopa or Levodopa or any of the excipients or any related drug.
2. History or presence of any disease or condition which might compromise the hemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal, or any other body system.
3. Ingestion of a medicine (prescribed & over the counter (OTC) medication including herbal remedies and MAO inhibitors) at any time within 30 days before first dosing in Period I. In any such case, subject selection will be at the discretion of the Principal Investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-10-29 (Actual); Primary Completion 2022-01-25 (Estimated); Study Completion 2022-03-25 (Estimated)

PRIMARY OUTCOMES:
Cmax of the pharmacokinetics of WD-1603 extended-release formulations and carbidopa and levodopa tablets 25mg/100mg from the morning of day 1 to the morning of day 2. | 24 hours-from morning of Day 1 to morning of Day 2
  To evaluate Cmax (Maximum Plasma Concentration) of the pharmacokinetics of WD-1603 extended-release formulations and carbidopa and levodopa tablets 25mg/100mg following three times a day after oral administration in fasting and fed conditions in healthy subjects.
The duration (hours) for the levodopa concentrations ≥ 50% of Cmax between WD-1603 extended-release formulations and carbidopa and levodopa tablets following three times a day orally administration in healthy subjects. | 24 hours-from morning of Day 1 to morning of Day 2
  To compare the duration (hours) for the levodopa concentrations ≥ 50% of Cmax, where maximum measured plasma concentration after 1st dose or 2nd or 3rd dose for each dose interval.

CONTACTS AND LOCATIONS:
Overall Officials: Akash Patel, M.D., Principal Investigator — Lambda Therapeutic Research Ltd.
Locations (1):
- Lambda Therapeutic Research Ltd., Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No